CLINICAL TRIAL: NCT00003552
Title: Phase I/II Study of HLA-Matched Peripheral Blood Mobilized Hematopoietic Progenitor Cell Transplantation Followed by Allogeneic T-cell Infusion as Adoptive Immunotherapy in Patients With Metastatic Melanoma
Brief Title: Chemotherapy and Peripheral Stem Cell Transplantation in Treating Patients With Metastatic Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066609; NHLBI-98-H-0006; NCT00001739 (obsolete NCT alias)
Record Dates: First submitted 2007-03-01; First posted 2007-03-05 (Estimated); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Stage IV Melanoma; Recurrent Melanoma
Keywords: adult solid tumor; body system/site cancer; cancer; melanoma; recurrent melanoma; skin tumor; solid tumor; stage IV melanoma; stage, melanoma
MeSH Terms: conditions — Melanoma; Neoplasms; Skin Neoplasms | interventions — Antilymphocyte Serum; Cyclophosphamide; fludarabine

INTERVENTIONS:
Drug: allogeneic lymphocytes
Drug: anti-thymocyte globulin
Drug: cyclophosphamide
Drug: fludarabine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Peripheral stem cell transplantation may allow doctors to give higher doses of chemotherapy and kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of chemotherapy plus peripheral stem cell transplantation in treating patients with metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Identify an antitumor effect of allogeneic peripheral blood stem cell transplantation (PBSCT) in patients with metastatic melanoma.

II. Evaluate the safety and toxicity of a nonmyeloablative, low intensity, preparative regimen followed by an HLA-matched allogeneic PBSCT in these patients.

III. Monitor engraftment by measuring donor-recipient chimerism in lymphoid and myeloid lineages in these patients.

IV. Investigate the relationship between donor-host chimerism and the incidence of acute and chronic graft-versus-host disease in this patient population.

V. Investigate the effect of lymphocyte infusions on donor-host chimerism in this patient population.

VI. Determine disease-free survival, overall survival, and mortality from the procedure or tumor progression in this patient population.

PROTOCOL OUTLINE: This is a dose-escalation study of a conditioning regimen. Patients receive 1 of 3 dose levels of chemotherapy prior to peripheral blood progenitor cell (PBPC) transplantation. Patients at dose level 1 receive cyclophosphamide IV over 1 hour on days -7 and -6 and fludarabine IV over 30 minutes daily on days -5 to -1. Patients at dose level 2 receive cyclophosphamide IV over 1 hour on days -7 and -6, fludarabine IV over 30 minutes daily on days -5 to -1, and antithymocyte globulin daily on days -5 to -2. Patients at dose level 3 receive cyclophosphamide IV over 1 hour daily on days -8 to -6, fludarabine IV over 30 minutes daily on days -5 to -1, and antithymocyte globulin daily on days -5 to -2.

Patients undergo mobilized CD34+ PBPC transplantation on day 0. PBPC transplantation may be repeated on days 1 and 2 if deemed necessary.

Patients with progressive disease on days 15-30, day 60, or day 100, without graft-versus-host disease, receive infusion(s) of donor lymphocytes. Further donor lymphocyte infusions after day 100 may be given at the discretion of the attending physician.

Patients are followed every 2 months for 6 months, every 3 months for the next 2 years, and then every 6 months until year 5 posttransplantation.

PROJECTED ACCRUAL:

A total of 40 patients will be accrued for this study.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Histologically confirmed metastatic melanoma not amenable to complete surgical resection and progressive despite immunotherapy and/or chemotherapy Bidimensionally evaluable clinically or radiographically HLA 6/6 or 5/6 matched sibling donor available No CNS metastases --Prior/Concurrent Therapy-- See Disease Characteristics At least 30 days since prior treatment for melanoma --Patient Characteristics-- Age: 18 to 60 Performance status: ECOG 0-1 Life expectancy: At least 3 months Hematopoietic: Not specified Hepatic: Bilirubin no greater than 4 mg/dL Transaminases no greater than 3 times upper limit of normal Renal: Creatinine no greater than 2.5 mg/dL Cardiovascular: Left ventricular ejection fraction greater than 40% Pulmonary: DLCO greater than 65% of predicted Other: HIV negative No major organ dysfunction precluding transplantation No other malignancies except basal cell or squamous cell skin cancer No psychiatric disorder or mental deficiency that would preclude study Not pregnant or nursing

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Dates: Start 1999-01; Study Completion 2002-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard W. Childs, Study Chair — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Heart, Lung, and Blood Institute, Bethesda, Maryland, United States